CLINICAL TRIAL: NCT05238376
Title: The Effect of High-intensity Interval Training (HIIT) and Resistance Training on Function, Health, and Quality of Life Outcomes Following Hematopoietic Stem Cell Transplant
Brief Title: Survivorship Post-HCT Optimization Program
Acronym: S-POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00110028
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Experimental): These are patients who are 90 (±30) days post-allogeneic hematopoietic stem cell transplant. Patients will complete 12 weeks of exercise training. Patients will also complete assessments to evaluate physical function, cognitive function, mental health, social support, nutrition and diet, symptoms, quality of life, and financial status. They will use devices to capture activity data and vital signs. They will collect bio-specimens to assess microbiota and biomarkers.
  Interventions: Behavioral: Exercise training
- Caregiver (Experimental): These are the assigned caregivers for the transplant patients. Caregivers will complete 12 weeks of exercise training. Caregivers will also complete assessments to evaluate physical function, caregiver support, and physical activity and exercise. They will collect bio-specimens to assess microbiota.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — 12 weeks of high intensity interval training (HIIT) (3x/week) and resistance training (2x/week)

SUMMARY:
The purpose of this project is to investigate the effects of 12 weeks of high-intensity interval training (HIIT) and resistance training on several domains of health including physical function, cognitive function, mental health, and quality of life in patients who have undergone hematopoietic stem cell transplant (HCT). In addition, the project will determine the effects of 12 weeks of HIIT and resistance training on physical function, caregiver strain, mental health, and caregiver confidence in individuals who are providing care for patients undergoing HCT.

ELIGIBILITY:
Patient Inclusion Criteria:

1. ≥18 years old
2. English speaking
3. Within 90 ± 30 days post allogenic HCT

Caregiver Inclusion Criteria:

1. ≥18 years old
2. English speaking
3. Providing post-discharge care for the patient who has undergone HCT

Patient and Caregiver Exclusion Criteria:

1. Have an absolute contraindication to exercise including a recent acute cardiac event (<6 months), unstable angina, uncontrolled dysthymias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspects or known dissecting aneurism, or coronary artery disease.
2. In addition to these absolute contraindications, the patient and caregiver will complete cardiopulmonary exercise testing (CPET) where the heart rate and heart rhythm will be monitored via a 12-lead ECG before, during, and after the test. The results from the CPET will be reviewed by a physician before the subject is cleared to participate in the HIIT and resistance training program. If the participant is not cleared by the physician following the CPET, then the patient and his or her caregiver will not be eligible to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed exercise program, as measured by number of total sessions completed | 12 weeks
Compliance to prescribed HIIT sessions, as measured by total session time (in minutes) | 12 weeks
Compliance to prescribed HIIT sessions, as measured by number of intervals completed | 12 weeks
Compliance to prescribed HIIT sessions, as measured by number/percentage of intervals meeting target heart rates | 12 weeks
Compliance to prescribed resistance sessions, as measured by number of sets completed | 12 weeks
Compliance to prescribed resistance sessions, as measured by number of repetitions completed | 12 weeks

SECONDARY OUTCOMES:
Change in physical function/activity, as measured by SPPB | Baseline, Post-intervention (week 12), 1 Year
  All the task points are added which make the SPPB score. The cut-point for the SPPB is a score of 10. The cumulative and sections scores are assessed individually and comprehensively. This assessment score will be used as a tool for evaluating lower extremity functioning in older persons.
Change in physical function/activity, as measured by 6-minute walk test | Baseline, Post-intervention (week 12), 1 Year
  The baseline for each patient is made through an algorithm that factors the patients age and gender. The patient's score is compared to what a person that is the patient's same age and gender would get. This comparison is then used as a tool to assess aerobic capacity or endurance.
Change in physical function/activity, as measured by 30-second sit-to-stand | Baseline, Post-intervention (week 12), 1 Year
  Subjects will sit in a chair with their arms crossed over their chest and rise to a standing position, then return to seated position. They will repeat this as many times as they can in 30 seconds.
Change in physical function/activity, as measured by grip strength | Baseline, Post-intervention (week 12), 1 Year
  The hand grip is an indicator of upper body strength and has been found to be a good predictor of future functional limitations and disabilities. The hand grip score is determined based on how quickly the participant can squeeze the hand dynamometer.
Change in physical function/activity, as measured by Fried Frailty | Baseline, Post-intervention (week 12), 1 Year
  The scores of all of the sections are added and if the patient has a score greater or equal to three this assessment deems that the patients is frail. If the patient has a score between 1-2 the patient is deemed pre-frail.
Change in physical function/activity, as measured by PROMIS Physical Function | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in physical function/activity, as measured by bioelectrical impedance (BIA) | Baseline, Post-intervention (week 12), 1 Year
  Participants will have body composition assessed by bioelectrical impedance spectroscopy (BIS) via a bioimpedance analysis (BIA) device. BIA equipment does not measure muscle mass directly, but instead derives an estimate of muscle mass based on whole-body electrical conductivity.
Change in physical function/activity, as measured by CPET | Baseline, Post-intervention (week 12), 1 Year
  Exercise capacity will be assessed using a symptom-limited Cardiopulmonary Exercise Test (CPET) on a cycle ergometer or for a six-minute step test with expired gas analysis to determine VO2peak, according to guidelines for clinical populations (Jones et al., 2012). All CPET data will be recorded as the highest 30-second value elicited during the CPET.
Change in physical function/activity, as measured by Intramuscular Adipose Tissue (IMAT) | Baseline, Post-intervention (week 12), 1 Year
  Longitudinal and transverse ultrasound images of the m. rectus femoris, vastus lateralis, m. intercostalis / m. pectoralis, (head) m. temporalis, and/or (head) styloglossus. Complex grayscale analysis of the images is used to calculate the IMAT.
Change in physical function/activity, as measured by Intramuscular Glycogen Content (IMGC) | Baseline, Post-intervention (week 12), 1 Year
  Longitudinal and transverse ultrasound images of the m. rectus femoris, vastus lateralis, m. intercostalis / m. pectoralis, (head) m. temporalis, and/or (head) styloglossus. Complex grayscale analysis of the images is used to calculate the IMGC.
Change in physical function/activity, as measured by muscle thickness | Baseline, Post-intervention (week 12), 1 Year
  Longitudinal and transverse ultrasound images of the m. rectus femoris, vastus lateralis, m. intercostalis / m. pectoralis, (head) m. temporalis, and/or (head) styloglossus, using greyscale analyses.
Change in physical function/activity, as measured by muscle area | Baseline, Post-intervention (week 12), 1 Year
  Longitudinal and transverse ultrasound images of the m. rectus femoris, vastus lateralis, m. intercostalis / m. pectoralis, (head) m. temporalis, and/or (head) styloglossus, using greyscale analyses.
Change in physical function/activity, as measured by subcutaneous fat layer thickness | Baseline, Post-intervention (week 12), 1 Year
  Longitudinal and transverse ultrasound images of the m. rectus femoris, vastus lateralis, m. intercostalis / m. pectoralis, (head) m. temporalis, and/or (head) styloglossus, using greyscale analyses.
Change in cognitive function, as measured by Montreal Cognitive Assessment (MOCA) | Baseline, Post-intervention (week 12), 1 Year
  This administered assessment is subdivided into visuospatial/executive (5pts), naming (3pts), memory (no points), attention(5pts), language(3pts), abstraction(2pts), delayed recall(5pts), and orientation(6pts). All the subdivided sections have as many questions as they have points. For analysis, the cut point is if the patient has less than 26 points.
Change in cognitive function, as measured by PROMIS Cognitive Function | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in cognitive function, as measured by RBANS | Baseline, Post-intervention (week 12), 1 Year
  RBANS evaluation produces five index scores as well as a total summary score, and total scaled score. Scores range from 40 to 160, with higher scores indicating better performance (Smith et al., 2014). The scaled score classifies neuropsychological performance as: extremely low (69 and below), borderline (70-79), low average (80-89), average (90-109), high average (110-119), superior (120-129), and very superior (130 and above) (Batty et al., 2016; Randolph et al., 1998).
Change in cognitive function, as measured by Trail making test | Baseline, Post-intervention (week 12), 1 Year
  Trail Making Test parts A and B (TMT-A and -B) will be used for identification of cognitively impairment. Total time to completion will be used as outcome variable for both parts (ranging from 0 to 300 seconds, with higher scores indicating worse performance (Smith et al., 2014). An adjusted mean T-score also will be calculated ranging from 0 to 100 (mean score 50, higher score indicating better performance). The T-score can be adjusted for age, sex, education and ethnicity.
Change in cognitive function, as measured by Brief Cope | Baseline, Post-intervention (week 12), 1 Year
  Scores are presented for three overarching coping styles as average scores (sum of item scores divided by number of items), indicating the degree to which the respondent has been engaging in that coping style.
Change in mental health, as measured by PHQ-9 | Baseline, Post-intervention (week 12), 1 Year
  The PHQ-9 consists of 9 items, each of which is scored 0 to 3, giving a 0 to 27 severity score
Change in mental health, as measured by PC-PTSD/PCL-5 | Baseline, Post-intervention (week 12), 1 Year
  PC-PTSD is a 5 item screen to identify patients with probable PTSD. If the patient screens positive, they then take the PCL-5. The PCL-5 is a 20 item screen to assess symptoms of PTSD.
Change in mental health, as measured by PROMIS Depression | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in mental health, as measured by PROMIS Anxiety | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in diet/nutrition, as measured by Perioperative Nutrition Screen (PONS) | Baseline, Post-intervention (week 12), 1 Year
  PONS analyzes BMI, weight loss, and food intake to screen for preoperative nutrition risk
Change in diet/nutrition, as measured by PG-SGA/Clinician SGA | Baseline, Post-intervention (week 12), 1 Year
  Scores for each section can range from 0-4 depending on severity and nutritional impact. The sum of all scores provides the Total PG-SGA score, which can be used to indicate the need for intervention (Bauer et al., 2002)
Change in diet/nutrition, as measured by ASA-24 | Baseline, Post-intervention (week 12), 1 Year
  ASA-24 is a self-administered 24-hour diet recall
Change in diet/nutrition, as measured by Food Security | Baseline, Post-intervention (week 12), 1 Year
  Participants will be given the USDA food security survey to review their food securities or insecurities. This is a 10 item survey.
Change in social support, as measured by PROMIS Emotional Support | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in social support, as measured by PROMIS Social Isolation | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in social support, as measured by Lorig Self Efficacy | Baseline, Post-intervention (week 12), 1 Year
  The Self-Efficacy to Manage Chronic Disease Scale is made up of 6-items on a visual analog scale, ranging from 1 (not at all confident) to 10 (totally confident).
Change in social support, as measured by CFC-14 | Baseline, Post-intervention (week 12), 1 Year
  CFC-14 is a 14 item questionnaire to assess a patient's consideration of immediate and consideration of future consequences
Change in social support, as measured by Brief Resilience Scale | Baseline, Post-intervention (week 12), 1 Year
  BRS assesses the patient's ability to recover from stress. The possible score range on the BRS is from 1 (low resilience) to 5 (high resilience).
Change in caregiver support, as measured by Caregiver Strain index | Baseline, Post-intervention (week 12), 1 Year
  Tool to assess strain on long-term caregivers
Change in caregiver support, as measured by Preparedness for Caregiving assessment | Baseline, Post-intervention (week 12), 1 Year
  Items are scored by calculating the mean of all items with a range of 0-4. The higher the score, the more prepared the caregiver feels to give care.
Change in caregiver support, as measured by FACT-GP | Baseline, Post-intervention (week 12), 1 Year
  21 item assessment scored on a 5-point Likert scale
Change in caregiver support, as measured by PHQ-2 | Baseline, Post-intervention (week 12), 1 Year
  The PHQ-9 consists of 2 items, each of which is scored 0 to 3, giving a 0 to 6 severity score
Change in caregiver support, as measured by PCL-5 | Baseline, Post-intervention (week 12), 1 Year
  The PCL-5 is a 20 item screen to assess symptoms of PTSD.
Change in caregiver support, as measured by Ego Resiliency | Baseline, Post-intervention (week 12), 1 Year
  14 item survey scored from 0-56, where a higher score indicates higher level of resiliency
Change in caregiver support, as measured by PROMIS Depression | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in caregiver support, as measured by PROMIS Anxiety | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in caregiver support, as measured by PROMIS Emotional Support | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in caregiver support, as measured by PROMIS Social Isolation | Baseline, Post-intervention (week 12), 1 Year
  The questions are asked as interval format with "0-Never" through "5-Always." Each of the PRO instruments will be scored on the T-score metric, where 50 is the mean of a reference population and 10 is the standard deviation of that population.
Change in microbiota diversity, as measured by skin swabs | Baseline, Post-intervention (week 12), 1 Year
  Skin swab samples batch sequenced and microbiome analyzed
Change in microbiota diversity, as measured by stool samples | Baseline, Post-intervention (week 12), 1 Year
  Changes in stool samples as measured by 16s rRNA sequencing
Change in biomarkers of inflammation and frailty, as measured by blood plasma samples | Baseline, Post-intervention (week 12), 1 Year
  Assays evaluating angiogenic, stromal, and inflammatory markers and markers of aging (the Pepper Panel) are used to assess inflammation and frailty
Overall survival, as measured by medical record review | 1 year
Disease-free survival, as measured by medical record review | 1 year
Rate of bacterial infection, as measured by medical record review | 1 year
Rate of fungal infection, as measured by medical record review | 1 year
Rate of viral infection, as measured by medical record review | 1 year
Rate of overall infection, as measured by medical record review | 1 year
Rate of hospital admission, as measured by medical record review | 1 year
Rate of intensive care unit admission, as measured by medical record review | 1 year
Hospital length of stay, as measured by medical record review | 1 year
Intensive care unit length of stay, as measured by medical record review | 1 year
Number of patients with grade 2+ graft-versus-host disease, as measured by medical record review | 1 year
Transplant length of stay (in days), as measured by medical record review | 1 year
Number of patients who returned to work, as assessed by Work Assessment | 1 year
Number of falls, as assessed by Falls questionnaire | 1 year
  Participants will answer Yes/No to whether they have had any falls in the preceding 6 months
Number of subjects who experienced delirium, as assessed by DOS assessment | 1 year
  The Delirium Observation Screening Scale is a 13-item observational scale of verbal and nonverbal behavior. The observations can be done during regular care. The DOS is used to optimize recognition of delirium.
Change in quality of life, as assessed by FACT-BMT assessment | Baseline, Post-intervention (12 weeks), 1 Year
  50 item assessment. Higher total and domain scores indicate greater quality of life.
Change in quality of life, as assessed by EQ-5D-5L assessment | Baseline, Post-intervention (12 weeks), 1 Year
  The 5D represents 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Five levels of severity are measured, as indicated by the "5L," ranging from "no problems" to "extreme problems." All scores are converted into a summary index.
Change in quality of life, as assessed by OARS IADL assessment | Baseline, Post-intervention (12 weeks), 1 Year
  OARS IADL is a 7 item assessment that asks what level of assistance is needed to do 7 different activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Chenyu Lin, MD, Principal Investigator — Duke University
Locations (1):
- Duke Adult Blood and Marrow Transplant Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No